CLINICAL TRIAL: NCT03090607
Title: A 12-month Double-blind, Randomized, Controlled Pivotal Trial to Evaluate the Safety and Efficacy of Endoluminal Aluvra™ for the Treatment of Gastroesophageal Reflux Disease
Brief Title: Novel Endoluminal Clinical TreAtment of Reflux
Acronym: NECTAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Impleo Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NECTAR
Record Dates: First submitted 2017-03-15; First posted 2017-03-27 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Aluvra™ (Experimental): Endoscopic injection of bulking agent (Aluvra) to the lower esophageal sphincter
  Interventions: Device: Aluvra™
- Saline (Sham Comparator): Endoscopic injection of saline
  Interventions: Drug: Saline

INTERVENTIONS:
Device: Aluvra™ — Endoscopic injection of bulking agent to the lower esophageal sphincter
  Other Names: injectable bulking agent for GERD
  Arms: Aluvra™
Drug: Saline — Endoscopic injection of saline
  Arms: Saline

SUMMARY:
This is a prospective, multi-center, double-blind, crossover, randomized controlled trial designed to demonstrate the safety and efficacy of Aluvra for the treatment of GERD.

ELIGIBILITY:
Inclusion Criteria:

1. History of heartburn-like pain, regurgitation, or both prior to the initiation of proton pump inhibitor (PPIs) therapy.
2. History of GERD symptoms of at least six months despite continuous PPIs.
3. GERD-HRQL score ≥15 after discontinuing PPI therapy.
4. GERD-HRQL score improvement of at least 6 points while on PPIs, with at least 4-point improvement in heartburn subscore.
5. A minimum GERD-HRQL score while on PPIs of 2.
6. Pathologic acid exposure time, a baseline pH <4.0 for ≥ 5.3% of time during a 48-hour evaluation period.
7. Twenty two years of age or older.
8. Life expectancy of at least two years.
9. Willing and able to return to the clinic or hospital for all evaluation procedures scheduled throughout the course of this study.
10. Is capable of understanding clinical study procedures and giving informed consent.

Exclusion Criteria:

1. Unable to tolerate an endoscopic procedure
2. Presence of esophageal or gastric varices
3. Presence of erosive esophagitis (LA Classification of C or D)
4. Presence of a hiatal hernia > 2 cm
5. Presence of Barrett's esophagus
6. Presence of esophageal motility disorder
7. History of or known esophageal stricture or gross esophageal anatomic abnormalities
8. Symptoms of dysphagia more than once per week within the last six months
9. Obesity (BMI ≥ 35)
10. Gastric or esophageal cancer undergoing active treatment
11. Received radiation therapy to the esophagus and has fibrosis of the tissue at the likely injection sites
12. Had an ablation procedure in the lower esophageal sphincter area
13. Has a condition that could lead to significant postoperative complications, including current infection, anticoagulant use, uncontrolled diabetes or autoimmune disorder
14. Enrolled in a concurrent clinical trial
15. Inability to comply with study protocol due to a chronic disease, psychiatric illness, alcoholism, drug abuse, or geographic distance (as determined by investigator)
16. Pregnant and/or given birth in the previous twelve months or who plan to become pregnant in the next twelve months
17. Prior gastric or GERD surgery

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Aluvra- GERD HRQL | 12 months
  Efficacy will be established through two co-primary objectives. The first co-primary endpoint will be to compare response rates between treatment group and control group at 12 months based on the GERD-Health Related Quality of Life questionnaire.
Efficacy of Aluvra- Esophageal PH | 12 months
  Efficacy will be established through two co-primary objectives. The second co-primary endpoint will be to compare change from baseline in total percent time esophageal pH <4 between the treatment group vs. the sham control group at 12 months.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Keck School of Medicine of USC, Los Angeles, California
  - Digestive Health Center, Palo Alto, California
  - SOFI - Center for Esophageal Wellness, Englewood, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - Esophageal Institute of Atlanta, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University in Saint Louis, St Louis, Missouri
  - The Oregon Clinic, Gastrointestinal and Minimally Invasive Surgery Division, Portland, Oregon
  - Aurora Medical Center Summit, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided